CLINICAL TRIAL: NCT06495177
Title: European Survey of Cardiovascular Disease Prevention, Diabetes and Chronic Kidney Disease
Brief Title: European Survey of Cardiovascular Disease Prevention, Diabetes and Chronic Kidney Disease (EUROASPIRE VI)
Acronym: EUROASPIRE VI
Status: Recruiting | Type: Observational
Sponsor: European Society of Cardiology (Network)
Collaborators: National Institute for Prevention and Cardiovascular Health, Ireland (Other)
Responsible Party: Sponsor
Other Study IDs: EAVI
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Coronary Disease; Acute Coronary Syndrome; Unstable Angina; ST Elevation Myocardial Infarction; Non-ST Elevation Myocardial Infarction
MeSH Terms: conditions — Coronary Disease; Acute Coronary Syndrome; Angina, Unstable; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hospital Arm: Patients presenting with coronary heart disease
- Primary Care Arm: People at high risk of cardiovascular disease

SUMMARY:
The goal of this observational study is to provide a unique European picture of preventive action by cardiologists, other specialists and primary care physicians looking after patients with coronary heart disease (CHD), individuals at high cardiovascular disease risk and all those with hypertension, dyslipidaemia (including familial hypercholesterolaemia), diabetes and dysglycaemia and chronic kidney disease (CKD) and determine whether the European guidelines on cardiovascular disease prevention, hypertension, lipids, diabetes and chronic kidney disease are being followed.

DETAILED DESCRIPTION:
EUROASPIRE is a multicentre European study in coronary patients and individuals at high risk of developing cardiovascular disease (CVD), describing their management through lifestyle and use of drug therapies and providing an objective assessment of clinical implementation of current scientific knowledge. Five EUROASPIRE surveys have been carried out by the European Society of Cardiology so far: EUROASPIRE I in 1995-1997 in nine countries, EUROASPIRE II in 1999- 2000 in 15 countries, EUROASPIRE III in 2006-2009 in 22 countries, EUROASPIRE IV in 2012-2015 in 26 countries and EUROASPIRE V in 2016-2018 in 27 countries.

This sixth EUROASPIRE survey will investigate the cardiometabolic and renal continuum in both secondary and primary cardiovascular disease prevention in 2023-2025 under the auspices of the European Society of Cardiology, Global Registries And Surveys Programme (GRASP). As in the previous EUROASPIRE surveys this survey will be focused on hospital patients with CHD, with and without diabetes mellitus, and apparently healthy individuals in primary care at high risk (hypertension, dyslipidaemia, diabetes) of developing CVD.

ELIGIBILITY:
Inclusion Criteria:

* Patients having signed an informed Consent
* Patients aged from 18 years old at the time of identification
* At least six and at most 24 months elapsed between the index event (the recruiting diagnostic or treatment criteria below) and the date of interview
* Patients meeting the recruiting diagnostic or treatment criteria:
* Coronary patients: Acute coronary events (acute coronary syndrome {STEMI or NSTEMI}, unstable angina) or an emergency or elective revascularisation for coronary artery disease (CABG, PCI)
* High cardiovascular disease (CVD) risk patients: patients free of CVD, who have been prescribed one or more of the following treatments: blood pressure and/or lipid-lowering and/or glucose lowering (diet and/or hypoglycaemic agents and/or insulin)

Exclusion Criteria:

* Patients living outside defined geographical areas
* Patients admitted to hospital from outside the geographical area or under the care of cardiologists in hospitals that do not participate in EUROASPIRE VI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is all consenting adult patients presenting with high risk of cardiovascular diseases identified by general practices medical note and all consenting adult patients presenting with coronary disease seen in clinic.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Proportions of hospital coronary patients and high risk individuals in primary care achieving European lifestyle, risk factors and therapeutic targets for cardiovascular disease prevention | 30 months
  The management of risk in terms of lifestyle intervention and the use of drug therapies will be evaluated in relation to the lifestyle and therapeutic goals defined in the national and European guidelines on cardiovascular disease prevention.

CONTACTS AND LOCATIONS:
Overall Officials: Pr David A Wood, MB ChB MSc, Study Chair — National Institute for Prevention and Cardiovascular Health; Pr John William McEvoy, MB BCh BAO MEd MHS PhD, Study Chair — National Institute for Prevention and Cardiovascular Health
Locations (1):
- Istanbul University, Cerrahpaşa Cardiology Institute, Istanbul, Turkey (Türkiye)